CLINICAL TRIAL: NCT03883425
Title: Frailty and Complexity Among Home Service Recipients: a Case-control Longitudinal Study
Brief Title: Frailty and Complexity Among Home Service Recipients
Acronym: fraXity
Status: Completed | Type: Observational
Sponsor: School of Health Sciences Geneva (Other)
Collaborators: Swiss National Science Foundation (Other); Geneva institution for homecare and assistance (imad) (Unknown)
Responsible Party: Principal Investigator, Catherine Ludwig, UAS associate professor, School of Health Sciences Geneva
Other Study IDs: AGP 84770
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Frail Elderly Syndrome
Keywords: Home Care Services; Geriatric Assessment; Aging; Frailty; Complexity; Nursing
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Case 1: formal home service recipients: Adults aged 65 or older living at home who receive formal home service (household, meal delivery, transportation, shopping) at least one a week
  Interventions: Other: interRAI-HC assessments
- Case 2: formal home care recipients: Adults aged 65 or older living at home who receive formal home care (shower/bath nursing assistance, nursing care) at least once a week
  Interventions: Other: interRAI-HC assessments
- Control: free of formal home care or home service: Adults aged 65 or older living at home who do not receive formal home care or home service.
  Interventions: Other: interRAI-HC assessments

INTERVENTIONS:
Other: interRAI-HC assessments — Standardized geriatric assessments done with the interRAI-HC instrument (Canadian French version 9.1) by trained nurses

SUMMARY:
The purpose of the study is to develop frailty and complexity computation algorithms based on the French version of the interRAI-HC and, in doing so, to provide homecare nurses with valid and reliable screening tools for their routine practice. By relying on a prospective observational case-control longitudinal study, the study intends to assess the predictive validity of the proposed indices with respect to undesirable health outcomes. Repeated measurement occasions, separated by 6-month intervals, will also allow for estimation of intra-individual change in frailty and complexity. In the study, elders living in the community and aged 65 or older are the target population, and three samples will be considered based on the a priori risks of adverse outcomes (case 1: formal home service recipients; case 2: formal home care recipients; control: free of formal home care or service). These groups will be compared on the observed rates of frailty and complexity and on their evolution over time. Results will allow for identification of subgroups of the aged population for whom early screening of frailty and complexity appears most relevant. Based on the findings, practice guideline will be proposed. They will entail the interpretation of the scores and recommendations for mounting adapted preventive strategies. Finally, the study will contribute to enhancing knowledge on the relation between frailty, a well-known concept in gerontology, and complexity, a concept increasingly referred to in the care literature but that still deserves operational and consensual definitions.

ELIGIBILITY:
Inclusion Criteria:

* living in the community (private home)
* resident of Canton Geneva, Switzerland
* ability to hold a conversation in French (expression, comprehension)
* oriented in time and space

Exclusion Criteria:

* living in hospital / nursing home
* not resident of Canton Geneva, Switzerland
* not fluent in French
* disoriented in time and space
* person under tutorship

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Community-dwelling older adults (aged 65 or older), fluent in French, living at home in Canton Geneva, Switzerland and volunteering to participate to the study.
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Frailty Index | at baseline
  Index with a value ranging from 0 to 100, computed as the sum of health deficits recorded with the interRAI-HC MDS divided by the number of deficits considered. Replication of Ludwig and Busnel, BMC, 2017 (REF2)
Complexity Index | at baseline
  Index with a value ranging from 0 to 100, computed as the sum of complexity items recorded with the interRAI-HC MDS divided by the number of items considered.
Change in frailty Index | at 6 months and at 12 months
  Change in the frailty index value; Expressed as a proportion, with the frailty index value at baseline as denominator and the observed frailty value as numerator.
Change in complexity Index | at 6 months and at 12 months
  Change in the complexity index value; Expressed as a proportion, with the complexity index value at baseline as denominator and the observed complexity value as numerator.

SECONDARY OUTCOMES:
Number of participants with falls | at 6 month, at 12 months
  Number of participants with falls in the 6 months prior each follow-up assessment (yes/no; if yes, number of falls that occurred); recorded prospectively by means of a life history calendar.
Number of participants with hospitalizations | at 6 month, at 12 months
  Number of participants with hospitalizations in the 6 months prior each follow-up assessment (yes/no; if yes, number of hospitalizations that occurred and lengths in days); recorded prospectively by means of a life history calendar.
Number of participants with physician visits | at 6 month, at 12 months
  Number of participants with physician visits in the 6 months prior each follow-up assessment (yes/no; if yes, number of visits that occurred); recorded prospectively by means of a life history calendar.
Number of participants with emergency admissions | at 6 month, at 12 months
  Number of participants with emergency admissions in the 6 months prior each follow-up assessment (yes/no; if yes, number of admissions that occurred); recorded prospectively by means of a life history calendar.
Mortality rate | at 6 month, at 12 months
  Number of deaths (yes/no); collected from relatives or through public databases (www.hommages.ch).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Ludwig, PhD, Principal Investigator — School of Health Sciences Geneva
Locations (1):
- School of Health Sciences Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data and analytical codes will be shared in the form of computerized data files in SPSS format (*.sav, *.sps). Variable specification are written in SPSS syntaxes (*.sps files). Syntaxes define for each variable (raw or recoded) its short name, its type (date, string, numerical), its label, its response values and labels, the values associated with missing data and the measurement scale. Whenever relevant, the syntax is annotated, providing, for example, the reference of the published guideline for recoding. All variable specifications are summarized in a codebook (generated by SPSS), which is completed by specifications on the data collection procedure and on the sources used as references for recoding. The dataset is free of individual personal information (named, dated of birth, addresses, etc.); unique numerical codes are used to identify participants.
Supporting Information: Study Protocol, Analytic Code
Time Frame: At the end of the study, the recoded data set (SPSS format, cleaned and coded), the data codebook, references for the measurement instruments and all other relevant information related to the project (e.g. protocol) will be deposited at DARIS/FORS for data sharing and reuse.
Access Criteria: Data access and reuse, as well as intellectual property rights issues will be addressed through FORS standard contractual arrangements for a) the conditions of data deposit and b) the conditions of data use by a third party.
URL: http://forscenter.ch

REFERENCES:
- [Background] Morris JN, Fries BE, Steel K, Ikegami N, Bernabei R, Carpenter GI, Gilgen R, Hirdes JP, Topinkova E. Comprehensive clinical assessment in community setting: applicability of the MDS-HC. J Am Geriatr Soc. 1997 Aug;45(8):1017-24. doi: 10.1111/j.1532-5415.1997.tb02975.x. PMID 9256857
- [Background] Ludwig C, Busnel C. Derivation of a frailty index from the resident assessment instrument - home care adapted for Switzerland: a study based on retrospective data analysis. BMC Geriatr. 2017 Sep 7;17(1):205. doi: 10.1186/s12877-017-0604-3. PMID 28882127
- [Derived] Busnel C, Vallet F, Ashikali EM, Ludwig C. Assessing multidimensional complexity in home care: congruencies and discrepancies between patients and nurses. BMC Nurs. 2022 Jun 24;21(1):166. doi: 10.1186/s12912-022-00942-x. PMID 35751082
- [Derived] Ludwig C, Busnel C. Protocol of a case-control longitudinal study (fraXity) assessing frailty and complexity among Swiss home service recipients using interRAI-HC assessments. BMC Geriatr. 2019 Aug 5;19(1):207. doi: 10.1186/s12877-019-1230-z. PMID 31382880